CLINICAL TRIAL: NCT03229785
Title: Determining Overall Improvement in the Quality of Life of Individuals Receiving Human Umbilical Cord Blood Plasma
Brief Title: Quality of Life Improvements With Cord Blood Plasma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hexagon Therapies, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HEXA0001
Record Dates: First submitted 2017-07-13; First posted 2017-07-26 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord Blood Plasma (Experimental): Six intravenous infusions of human umbilical cord blood plasma (HUCBP) during a twelve month study period. The amount of HUCBP being infused on each occasion is 50 mL.
  Interventions: Biological: Human Umbilical Cord Blood Plasma

INTERVENTIONS:
Biological: Human Umbilical Cord Blood Plasma — Plasma collected from human umbilical cord blood

SUMMARY:
This study aims to look at whether human umbilical cord blood plasma (HUCBP) is safe for intravascular (iv) administration; and whether it provides any reversal of frailty or other age-related biological measures.

DETAILED DESCRIPTION:
Participants that take part in this experimental treatment will receive six HUCBP infusions over a six month period, with a final check-up occuring six months after the last infusion. Blood samples will be collected before receiving each HUCBP infusion, and at the last check-up. Participants will also be asked to complete a medical questionnaire (SF 36) prior to the first infusion, and prior to each subsequent infusion. The medical questionnaire is four (4) pages in length and includes comprehensive questions about previous medical health and history.

Participation in the experimental treatment will involve monitoring by the Principal Doctor for a period of twelve months after the initial infusion of HUCBP. A second infusion is planned for one month after the initial infusion, a third infusion is planned for two months after the initial infusion, a fourth infusion is planned for three months after the initial infusion, a fifth infusion is planned for four months after the initial infusion,and a sixth infusion is planned for five months after the initial infusion. Participants will be asked to undergo the same blood tests and physical examinations performed at the time of the initial infusion at each of the five subsequent infusions (i.e. at one, two, three, four, and five months after the initial infusion). Twelve months after the initial infusion participants will be asked to attend for final blood tests and physical examinations. There will be no HUCBP infusion at the twelve-month visit.

Assessment criteria for the study include: (1) Short Form (36) Health Survey (SF 36); (2) Biomarkers of inflammation, oxidative stress, and growth factors; (3) Adrenal cortical hormone levels; (4) Telomere length; (5) Hand grip strength; (6) Body fat measurement; (7) DNA damage; and (8) Overall safety of intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or older
* Be willing and able to participate during the 12 month research period
* Women - must be diagnosed with infertility or menopause

Exclusion Criteria:

* Unable to perform tasks required for analysis of end points
* History of being hospitalized dues to infectious disease, such as pneumonia, within the last year
* Recent and current use of immunosuppressive drugs or HIV patients
* Scheduled to receive organ transplant
* Dementia or clinically relevant cognitive impairment
* Participants of previous (within 1 month) or current clinical trials
* Severe heart and kidney failure
* History of alcohol or drug abuse
* Known or suspected pregnancy
* Chronic Hepatitis B or C
* Diagnosis of cancer within 5 year of the study, or the possibility to contract cancer
* Anticancer chemotherapy and radiation therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
The Short Form (36) Health Survey (SF 36) | The investigators will determine changes in SF 36 scores collected at baseline and at 1 month after HUCBP infusion.
  SF 36 as a measure quality of life improvements compared to baseline

SECONDARY OUTCOMES:
Biomarkers of inflammation and oxidative stress. | Blood samples will be collected the day before the first infusion and 1 month after HUCBP infusion
  Blood samples will be tested for changes in biomarkers - compared to baseline measurements.
Adrenal cortical hormone levels as a measure of efficacy for anti-aging effects. | Testing will occur using blood samples that will be collected the day before the first infusion and 1 month after HUCBP infusion
  Blood samples will be tested for changes in adrenal cortical hormone as compared to the baseline measurements.
Telomere length as a measure of efficacy for anti-aging effects. | Testing will occur using blood samples that will be collected the day before the first infusion and 1 month after HUCBP infusion
  Blood samples will be tested for changes in the length of the telomere as compared to the baseline measurements (in particular, the investigators will be looking to see if HUCBP infusion protects telomere from shortening).
Hand grip strength as metric of anti-aging effects | Each participant will perform the grip strength test on the day of the first infusion (baseline) and 1 month after HUCBP infusion
  Hand grip strength will be tested on the day of the initial infusion and 1 month after HUCBP infusion. The investigators will assess changes in handgrip strength compared to the baseline, collected on the day of the first infusion.
Body fat measurements | Body fat measurements of each participant will occur one day before the first infusion and 1 month after HUCBP infusion
  Baseline body-fat measurements will be taken on the day of the first HUCBP infusion using calipers. These measurements will be compared to additional measurements collected 1 month after HUCBP infusion. The investigators will assess changes in body-fat measurements compared to baseline.
Extent of DNA damage as a measure of efficacy for anti-aging effects | White blood cells isolated from blood samples collected the day before the first infusion and 1 month after HUCBP infusion.
  Blood samples will be tested to assess changes of 8-hydroxyguanine (a common marker of DNA damage) in whole blood - compared to baseline measurements.

IPD SHARING:
Plan to Share IPD: No